CLINICAL TRIAL: NCT07028333
Title: Effects of Different Dual-Task Exercises on Motor and Cognitive Functions in Children With Mild Mental Retardation
Brief Title: Effects of Different Dual-Task Exercises in Children With Mild Mental Retardation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melike Nur AKGÖĞ, Master's Degree Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUCAkgog001
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Mental Retardation
Keywords: Dual-Task Exercise; Motor Function; Cognitive Function; Rehabilitation; mental retardation; Balance; physiotherapy and Rehabilitation
MeSH Terms: conditions — Intellectual Disability | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a three-arm, randomized controlled trial involving children aged 8-12 with mild mental retardation. Participants will be randomly assigned to one of three groups: Motor-Motor Dual Task Exercise, Motor-Cognitive Dual Task Exercise, or Control.
  The Motor-Motor group will perform walking and balance exercises combined with motor tasks under physiotherapist supervision. The Motor-Cognitive group will perform the same physical exercises combined with cognitive tasks. The Control group will follow standard walking and balance exercises at home, monitored by parents.
  Interventions will last six weeks, conducted twice a week for about 40 minutes per session. Assessments of motor function, cognitive performance, and quality of life will be conducted before and after the intervention by blinded evaluators. Data will be analyzed to compare group outcomes and determine the effects of dual-task exercises on motor and cognitive functions in children with mild mental re
Masking Description: his study is a three-arm, randomized controlled interventional trial involving children aged 8-12 with mild mental retardation. Participants will be randomly assigned to one of three groups: Motor-Motor Dual Task Exercise, Motor-Cognitive Dual Task Exercise, or Control.
  The Motor-Motor group will perform walking and balance exercises combined with motor tasks under physiotherapist supervision. The Motor-Cognitive group will perform the same physical exercises combined with cognitive tasks. The Control group will follow standard walking and balance exercises at home, monitored by parents.
  Interventions will last six weeks, conducted twice a week for about 40 minutes per session. Assessments of motor function, cognitive performance, and quality of life will be conducted before and after the intervention by blinded evaluators. Data will be analyzed to compare group outcomes and determine the effects of dual-task exercises on motor and cognitive functions in children with mild mental ret
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- motor-motor dual task exercise group (Experimental): While this group performs walking and balance exercises accompanied by a physiotherapist, it will perform motor tasks.
  Interventions: Behavioral: Motor-Motor Dual Task Exercise Group
- Motor-Cognitive Dual Task Exercise Group (Experimental): While this group performs walking and balance exercises accompanied by a physiotherapist, it will perform cognitive tasks.
  Interventions: Behavioral: Motor-Cognitive Dual Task Exercise Group
- Control Group (Placebo Comparator): Standard walking and balance exercises will be given to the control group at home and followed by parents.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Motor-Motor Dual Task Exercise Group — Participants in this group will perform motor tasks (such as ball handling, throwing, holding) accompanied by physiotherapist. Exercises will last about 40 minutes, 2 days a week, 6 weeks.
  Arms: motor-motor dual task exercise group
Behavioral: Motor-Cognitive Dual Task Exercise Group — This group will also do walking and balance exercises with the physiotherapist, while simultaneously doing cognitive tasks (rhythmic counting, saying color names, finding words, etc.). The exercises will last approximately 40 minutes, 2 days a week, for 6 weeks.
  Arms: Motor-Cognitive Dual Task Exercise Group
Behavioral: Control Group — Standard walking and balance exercises will be given to the control group at home and followed by parents. Exercises will last about 40 minutes, 2 days a week, 6 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the effects of motor-motor and motor-cognitive dual-task exercises applied to children with mild mental retardation on their functional mobility, balance, cognitive function, and quality of life.

DETAILED DESCRIPTION:
Physical activity is a cornerstone of health and social well-being across all age groups. It holds significant physical, psychological, and social importance throughout an individual's life. Particularly in childhood, physical activity plays a critical role in shaping growth and development, enhancing cognitive functions, and establishing healthy habits that persist into adulthood. The World Health Organization (WHO) emphasizes the importance of physical activity for all age groups, highlighting its positive effects on children's cardiorespiratory fitness, muscle strength, bone health, mental health, cognitive functions, academic performance, and obesity prevention.

Children with mental retardation exhibit developmental delays across multiple domains compared to their typically developing peers. Mental retardation not only affects language, comprehension, learning, and socialization skills but also impairs motor abilities. These motor deficits contribute to reduced physical activity levels, increased sedentary behavior, and associated physical and psychological problems, which further restrict motor skill development. This cyclical relationship among mental retardation, motor function, and physical inactivity leads to decreased functionality, balance, strength, endurance, fitness, and flexibility. Consequently, children with mental retardation face challenges in daily activities and reduced quality of life.

In order to address these challenges, it is essential to implement exercise programs that target cognitive, social, and physical development in children with mental retardation. Performing daily movements often requires simultaneous execution of motor and cognitive tasks, known as dual-task activities. However, mental retardation significantly impairs the ability to perform such dual tasks. Existing literature indicates that dual-task interventions can improve balance, functional mobility, gait, and cognitive performance.

The current study aims to investigate the effects of dual-task exercise programs on motor and cognitive functions in children with mild mental retardation. Specifically, it examines whether motor-motor and motor-cognitive dual-task exercises improve these functions compared to a control group receiving standard walking and balance exercises. The intervention will be conducted over six weeks, with assessments performed before and after the program to measure motor skills, cognitive function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining parental consent
* Having an Intelligence Quotient between 51-70
* Having an educational diagnosis of mild mental retardation
* Being between the ages of 8-12
* Ability to understand Turkish instructions
* Ability to follow commands during the exercise program
* No additional disabilities that would prevent participation in the program

Exclusion Criteria:

* Having a metabolic or systemic disease
* Engaging in regular physical exercise
* Having visual or hearing impairments
* Presence of any condition that would interfere with compliance to assessment parameters

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 6 weeks
  The Pediatric Balance Scale (PBS), used to assess functional balance in children during daily activities, is a highly reliable measurement tool. It is an adapted version of the Berg Balance Scale specifically designed for children. The scale consists of 14 items evaluating functional movements such as standing up, picking up an object from the floor, transferring, balancing on one foot, and sitting. Each item is scored on a scale from 0 to 4, with 4 indicating the ability to perform the task independently. The maximum score is 56. Scores between 0-20 indicate poor balance, 21-40 indicate acceptable balance, and 41-56 indicate good balance.
Timed Up and Go Test | 6 weeks
  Description: The Timed Up and Go Test (TUG) is used to assess functional mobility by measuring walking speed, postural control, and balance. The test involves standing up from a standard-height chair without armrests, walking a distance of 3 meters, turning around, walking back to the chair, and sitting down. Participants perform one practice trial followed by three test trials, with the average time recorded in seconds. A shorter duration indicates better functional mobility and balance.
Tandem Walking Test | 6 weeks
  Description: The Tandem Walking Test is used to assess dynamic balance, a function primarily controlled by the cerebellum. Participants are instructed to walk 10 steps in a straight line, placing the heel of one foot directly in front of the toes of the other foot with each step, minimizing the base of support. The time taken to complete the 10 steps is recorded, and a shorter time indicates better dynamic balance.
Stroop Test | 6 weeks
  Description: The Stroop Test is a neuropsychological assessment that measures cognitive processing speed, selective attention, response inhibition, and cognitive flexibility-functions associated with the frontal lobe. It includes four cards, each containing six rows with four items per row. Participants are required to name the color of the ink used rather than the word itself, evaluating their ability to inhibit habitual responses and adapt to cognitive interference.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | 6 weeks
  The Pediatric Quality of Life Inventory (PedsQL), developed by Varni et al., is a validated tool used to assess health-related quality of life in children aged 2 to 18. The scale consists of four subdomains: physical, emotional, social, and school functioning. It provides a total score, a physical health summary score, and a psychosocial health summary score (derived from emotional, social, and school subscales). Each item is scored on a 5-point Likert scale, then transformed into a 0-100 scale, where higher scores indicate better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Melike N AKGÖĞ, MScStudent, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to privacy concerns and the sensitive nature of the data involving children with mild mental retardation. Additionally, sharing may be restricted to protect participant confidentiality and comply with ethical approvals. Data may be made available upon reasonable request and after necessary approvals to qualified researchers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT07028333/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT07028333/ICF_001.pdf